CLINICAL TRIAL: NCT00828880
Title: Restoration of Disk Height Through Non-Invasive Spinal Decompression is Associated With Decreased Discogenic Low-Back Pain: A Retrospective Cohort Study
Brief Title: Restoration of Disc Height Reduces Chronic Low Back Pain
Status: Completed | Type: Observational
Sponsor: NEMA Research, Inc. (Industry)
Collaborators: Axiom Worldwide, LLC (Industry)
Responsible Party: Joseph V. Pergolizzi, Jr., MD, NEMA Research, Inc
Other Study IDs: R-AXW01
Record Dates: First submitted 2009-01-22; First posted 2009-01-26 (Estimated); Last update posted 2009-01-26 (Estimated); Status verified 2009-01

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DRX9000
  Interventions: Device: DRX9000

INTERVENTIONS:
Device: DRX9000 — DRX9000 - non-invasive spinal decompression. Treatments 28 min 5 x/wk x 2wks, 3x/wk x 2 wks, 2x/wk x 2 wks for a total of 20 treatments in a 6-week period

SUMMARY:
The investigators hypothesize that a 6-week treatment of non-invasive spinal decompression reduces discogenic low back pain (LBP), increases lumbar disk height, and that an increase in lumbar disc height is associated with decreased LBP.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age;
* consented for the 6 weeks treatment protocol;
* presented with discogenic low back pain of at least 3 out of 10; AND
* current CT scan not older than 2 months.

Exclusion Criteria:

* metastatic cancer;
* previous spinal fusion or placement of stabilization hardware;
* instrumentation or artificial discs;
* neurologic motor deficits, bladder, or sexual dysfunction;
* alcohol or drug abuse; OR
* litigation for a health-related claim (in process or pending for workers' compensation or personal injury).

Limitations of the spinal decompression system also led to the exclusion of patients with extremes of height (< 147 cm or > 203 cm) and body weight (> 136 kg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Upper Valley Interventional Radiology, McAllen, Texas, United States

REFERENCES:
- [Derived] Apfel CC, Cakmakkaya OS, Martin W, Richmond C, Macario A, George E, Schaefer M, Pergolizzi JV. Restoration of disk height through non-surgical spinal decompression is associated with decreased discogenic low back pain: a retrospective cohort study. BMC Musculoskelet Disord. 2010 Jul 8;11:155. doi: 10.1186/1471-2474-11-155. PMID 20615252